CLINICAL TRIAL: NCT03840057
Title: Metoclopramide, Azithromycin, or Nondrug Pretreatment for Upper Gastrointestinal Bleeding to Reduce Second Endoscopy
Brief Title: Metoclopramide, Azithromycin, or Nondrug Pretreatment for UGIB to Reduce Second Endoscopy
Acronym: MANPURSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Waihong Chung (Other)
Responsible Party: Sponsor-Investigator, Waihong Chung, Fellow, Lifespan
Organization: Lifespan (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Gastro Intestinal Bleeding; Upper Gastrointestinal Bleeding
Keywords: GIB; UGIB
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Azithromycin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is comprised of two intervention arms, namely the azithromycin arm and the metoclopramide arm, as well as one placebo arm. The two interventions would be studied sequentially in order to simplify the logistical challenges of the blinding and placebo-control processes. The current study is comprised to two parts. During Part 1 of the study, participants are randomized to either azithromycin 500mg intravenous infusion or equivalent volume of 0.9% sodium chloride infusion in a 2-to-1 ratio. During Part 2 of the study, participants are randomized to either metoclopramide 10mg intravenous injection or equivalent volume of 0.9% sodium chloride injection in a 2-to-1 ratio. The 0.9% sodium chloride arm from the two parts of the study are pooled together to form the placebo arm during final analysis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Initial management of UGIB would be performed by the primary team without interference from the investigator. If a gastroenterology consult were placed by the primary team, the endoscopist on-call would evaluate the patient per routine care. If an early endoscopy is deemed appropriate and necessary based on the patient's clinical status, the participant is registered to a central electronic database, which would assign participants to the intervention arm or the placebo arm using a permuted block randomization process. The appropriate medication or placebo is prepared and distributed by the central inpatient pharmacy. The investigator, the endoscopist, the study participant, and the primary team are all blinded to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Azithromycin (Experimental): Participants randomized to the azithromycin arm would receive 250mL of reconstituted solution containing 500mg of generic azithromycin to be administered as a slow intravenous infusion over 1 hour by the primary team 30-120 minutes prior to endoscopy. No dosage adjustment is made for those with hepatic or renal impairment. No dose adjustment is made for geriatric population.
  Interventions: Drug: Azithromycin Injection
- Metoclopramide (Experimental): Participants randomized to the metoclopramide arm would receive 2mL of solution containing 10mg of generic metoclopramide to be administered as a direct intravenous push by the primary team 5-60 minutes prior to endoscopy. No dosage adjustment is made for those with hepatic impairment. A 50% dose reduction is made for those with creatinine clearance of less than 40mL/minute. No dose adjustment is made for geriatric population.
  Interventions: Drug: Metoclopramide Injectable Solution
- Placebo (Placebo Comparator): Participants randomized to the placebo arm during Part 1 (azithromycin) of the study would receive 250mL of 0.9% sodium chloride solution to be administered as a slow intravenous infusion over 1 hour by the primary team 30-120 minutes prior to endoscopy. Participants randomized to the placebo arm during Part 2 (metoclopramide) of the current study would receive 2mL of 0.9% sodium chloride solution to be administered as a direct intravenous push by the primary team 5-60 minutes prior to endoscopy.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Azithromycin Injection — Azithromycin, a semi-synthetic macrolide antibiotic derived from erythromycin. The role of azithromycin as a prokinetic agent was first reported in a retrospective cohort study, which showed azithromycin to be equivalent to erythromycin in accelerating gastric emptying in patients with gastroparesis. The aim of this intervention arm is to evaluate the effectiveness of azithromycin as a prokinetic agent in the management of UGIB.
  Arms: Azithromycin
Drug: Metoclopramide Injectable Solution — Metoclopramide, a 5-HT4 agonist and a dopamine D2-receptor antagonist, is approved for short-term treatment of gastroparesis. The use of metoclopramide as a prokinetic agent in the setting of UGIB has been previously studied, but the number of subject involved was too low to adequately power the studies. The aim of this intervention arm is to further evaluate the effectiveness of metoclopramide as a prokinetic agent in the management of UGIB.
  Arms: Metoclopramide
Drug: Sodium chloride 0.9% — Normal saline is used as a placebo control.
  Arms: Placebo

SUMMARY:
Early endoscopy is an integral part of the management plan for patients presenting with clinical signs of severe or ongoing UGIB. An accurate endoscopic diagnosis and successful endoscopic hemostasis is highly dependent on adequate visualization of the entire gastric mucosa. Metoclopramide has previously been investigated as a prokinetic agent to aid gastric emptying prior to endoscopy, but its widespread adoption is limited by a lack of high quality clinical evidence as well as concerns regarding side effects. Erythromycin is currently the only prokinetic agent recommended by the American and the European guidelines for use in selected patients in order to reduce the need for second endoscopy. Its clinical application, however, is limited by risk of arrhythmia, significant drug interactions, and frequent drug shortages. Azithromycin is structurally related to erythromycin, but is devoid of most adverse side effects associated with erythromycin use. Early evidence suggests that azithromycin may be an effective alternative to erythromycin in the treatment of gastroparesis. The current study, an interventional, randomized, triple-blinded, placebo-controlled clinical trial, is primarily aimed to evaluate the effectiveness of azithromycin as a prokinetic agent in the management of UGIB. It is also aimed to further evaluate the role of metoclopramide as a prokinetic agent in this setting. Outcome measures to be collected in this study include the need for secondary endoscopy, overall mortality, transfusion requirement, length of stay, requirement for surgery, and incidence of adverse side effects. Results from this study would help identify a safe, effective, and readily available prokinetic agent to be used prior to endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients ≥ 18 years of age at the time of presentation;
* 2. Admitted to Rhode Island Hospital (RIH) emergency room or inpatient services;
* 3. Presented with hematemesis, coffee ground emesis, or melena;
* 4. Upper endoscopy is planned within 24 hours of presentation or onset of bleeding.

Exclusion Criteria:

* 1. Known anaphylactic allergic reaction to erythromycin, azithromycin, and/or metoclopramide;
* 2. Concurrent use of certain medications associated with tardive dyskinesia (TD):
* a. Fluphenazine,
* b. Haloperidol,
* c. Loxapine,
* d. Paliperidone,
* e. Perphenazine,
* f. Pimozide,
* g. Risperidone,
* h. Thiothixene,
* i. Trifluoperazine;
* 3. Concurrent use of certain medications associated with torsade de pointes:
* a. Amiodarone,
* b. Chlorpromazine,
* c. Disopyramide,
* d. Dofetilide,
* e. Methadone,
* f. Procainamide,
* g. Quinidine,
* h. Sotalol;
* 4. Known history of TD, ventricular arrhythmias , or long QT syndrome;
* 5. Already received erythromycin and/or azithromycin within the past 10 days, or metoclopramide within the past 4 days for other indications;
* 6. Recipient of hematopoietic stem cell transplant;
* 7. History of Neisseria gonorrhoeae infection;
* 8. Pregnancy;
* 9. Prior gastrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Reduction in the Need for Second Endoscopy | 48 hours
  The primary outcome measure of effectiveness is a reduction in the need for second endoscopy within 48 hours of the first endoscopy. This primary outcome measure is chosen because it represents the basis of current American and European guideline recommendations regarding erythromycin.
Adverse Cardiac Side Effects related to Intervention | 5 days
  The primary cardiac outcome measure is the incidence of unstable arrhythmia, occurring within 5 days of azithromycin administration, requiring cardioversion or resulting in cardiac arrest.
Adverse Infectious Disease Side Effects related to Intervention | 30 days
  The primary infectious disease outcome measure is the incidence of C. difficile infection, occurring within 30 days of azithromycin administration.
Adverse Neurological Side Effects related to Intervention | 48 hours
  The primary neurological outcome measure is the incidence of any reversible or irreversible extrapyramidal symptom, such as acute dystonic reactions, akathisia, drug-induced Parkinsonism, and tardive dyskinesia, within 48 hours of metoclopramide administration.

SECONDARY OUTCOMES:
Quality of Endoscopic Visualization | 48 hours
  Endoscopic visibility is graded using the standard 4-point objective scoring system as described in most endoscopy literature. The corpus, fundus, and duodenal bulb are scored separately based on an independent review of the images captured by the endoscopist. If a second endoscopy is performed within 48 hours of the initial endoscopy, the presence of clinically significant lesions not identified during the first endoscopy is also measured.
All-Cause Mortality | 30 days.
  All-Cause Mortality within 30 days.
Number of Unit of Transfusion | 30 days
  Number of units of packed red blood cells transfused before hemostasis has been achieved or death.
Length of Hospital Stay | 30 days
  Length of hospital stay since admission for current episode of GIB.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gralnek IM, Dumonceau JM, Kuipers EJ, Lanas A, Sanders DS, Kurien M, Rotondano G, Hucl T, Dinis-Ribeiro M, Marmo R, Racz I, Arezzo A, Hoffmann RT, Lesur G, de Franchis R, Aabakken L, Veitch A, Radaelli F, Salgueiro P, Cardoso R, Maia L, Zullo A, Cipolletta L, Hassan C. Diagnosis and management of nonvariceal upper gastrointestinal hemorrhage: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Oct;47(10):a1-46. doi: 10.1055/s-0034-1393172. Epub 2015 Sep 29. PMID 26417980
- [Background] Laine L, Jensen DM. Management of patients with ulcer bleeding. Am J Gastroenterol. 2012 Mar;107(3):345-60; quiz 361. doi: 10.1038/ajg.2011.480. Epub 2012 Feb 7. PMID 22310222
- [Background] Lee A, Kuo B. Metoclopramide in the treatment of diabetic gastroparesis. Expert Rev Endocrinol Metab. 2010;5(5):653-662. doi: 10.1586/eem.10.41. PMID 21278804
- [Background] Larson JM, Tavakkoli A, Drane WE, Toskes PP, Moshiree B. Advantages of azithromycin over erythromycin in improving the gastric emptying half-time in adult patients with gastroparesis. J Neurogastroenterol Motil. 2010 Oct;16(4):407-13. doi: 10.5056/jnm.2010.16.4.407. Epub 2010 Oct 30. PMID 21103422
- [Background] Moshiree B, McDonald R, Hou W, Toskes PP. Comparison of the effect of azithromycin versus erythromycin on antroduodenal pressure profiles of patients with chronic functional gastrointestinal pain and gastroparesis. Dig Dis Sci. 2010 Mar;55(3):675-83. doi: 10.1007/s10620-009-1038-3. PMID 19924535
- [Background] Chini P, Toskes PP, Waseem S, Hou W, McDonald R, Moshiree B. Effect of azithromycin on small bowel motility in patients with gastrointestinal dysmotility. Scand J Gastroenterol. 2012 Apr;47(4):422-7. doi: 10.3109/00365521.2012.654402. Epub 2012 Feb 27. PMID 22364597